CLINICAL TRIAL: NCT00244218
Title: Response to Phenylketonuria to Tetrahydrobiopterin (BH4)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The FDA has approved Kuvan (BH4) as a therapeutic agent for phenylketonuria
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 01-269; FD-R-002600-01
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2015-06

CONDITIONS: Phenylketonuria
Keywords: phenylketonuria; hyperphenylalaninemia
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): Drug: tetrahydrobiopterin (BH4) Either placebo or BH4, 10mg/kg/day will be given for three months. Then the patient will be given three additional months of open label BH4 at the same rate.
  Interventions: Drug: tetrahydrobiopterin (BH4)
- Control Arm (Placebo Comparator): Drug: tetrahydrobiopterin (BH4) Either placebo or BH4, 10mg/kg/day will be given for three months. Then the patient will be given three additional months of open label BH4 at the same rate.
  Interventions: Drug: tetrahydrobiopterin (BH4)

INTERVENTIONS:
Drug: tetrahydrobiopterin (BH4) — Either placebo or tetrahydrobiopterin (BH4) , 10mg/kg/day will be given for three months. Then the patient will be given three additional months of open label BH4 at the same rate.
  Other Names: BH4

SUMMARY:
The purpose of this study is to determine whether tetrahydrobiopterin (BH4)is effective in treating patients with PKU.

DETAILED DESCRIPTION:
Phenylketonuria(PKU) is an autosomal recessive disorder caused by a defect in the enzyme phenylalanine hydroxylase(PAH). this incidence of PKU in the US is about 1:15,000 births. The disease is pan ethnic with more prevalence among individuals of European ancestry. Recently, a number of patients with PKU showed a marked decrease in their blood Phe levels when the cofactor for PAH, tetrahydrobiopterin (BH4) was given orally. All these patients had mutations in PAH while the metabolism of BH4 was normal. These observations were confirmed by several centers including a pilot study conducted in our institutions. In the study in our centers, we have identified 21 of 36 patients tested who responded favorably to BH4.

Recognizing the difficulties with phenylalanine restricted diet, an NIH Consensus Conference on PKU held in 1999, encouraged exploring different modalities for treating PKU, and BH4 is among these modalities. This proposal is a three year, double blind placebo control, multi-center study. An oral load of 10 mg/kg BH4 wil be given to patients with PKU to identify those that respond with lowering of blood Phe greater or equal to 30%. Blood Phe, tyrosine and dietary intake will be determined at zero time and 24 hours post load. From this group of BH4 responsive individuals, thirty-six will be enrolled in the double blind study. subjects will be randomized to the treatment of placebo group. Those who enter the trial will have zero time assessments including blood Phe and tyrosine, dietary intake, physical exam, kidney function, liver function and complete blood count (CBC). Phe and tyrosine and diet intakes, two prior to the study and the zero time, will be averaged and used as the baseline measures.

The subjects will be assigned randomly to take either 10mg/kg of BH4 orally or a placebo without BH4. Blood Phe, tyrosine and dietary intake will be obtained every other week throughout the 12 week study period. Liver function and kidney function and CBC's will be obtained monthly. Side effects will be evaluated and noted. Subjects will be instructed to record two day diet diaries prior to blood Phe sampling throughout the study. The NIH Consensus Report suggests maintaining blood Phe< 36 umol/l when less than 12 years of age or up to 900 umol/l after 12 years of age. These levels will be used to determine the efficacy end points of the study. At the end of three months, blood Phe and tyrosine, dietary intake, physical exam, kidney function, liver function and CBC will be performed. At this time efficacy of BH4 will be determined and all subjects will continue in an open label 12 weeks BH4 treatment, (10mg/kg/day), with assessments collected as in the first phase of the study. After the subject has had both phases they will be followed for an additional 3 months. The additional 3 month trial on BH4 will provide long term safety data from 18 subjects who took BH4 in both the first and second phase in a continuous fashion.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent or guardian must be capable of understanding and providing written informed consent
* Subjects must have Phenylketonuria (PKU)or hyperphenylalaninemia (HPA), defined as baseline blood Phe levels of >600 umol/L
* Subjects must be at least 10 years of age, and may be of either gender and any ethnic group
* Female subjects of childbearing potential must agree to use adequate birth control or refrain from sexual activity throughout study participation

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding
* Subjects who have concurrent diseases or conditions that require medication or treatment
* Subjects who require concomitant treatment with any drug known to inhibit folate synthesis
* Subjects who have been treated with any investigational drug within 30 days

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-04; Primary Completion 2009-03 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Blood Phe level decrease by 30% | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Matalon, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States